CLINICAL TRIAL: NCT05676112
Title: Safety of Nintedanib in Real World in China: a Non-interventional Study Based on Idiopathic Pulmonary (Interstitial) Fibrosis Registry China Study (PORTRAY) Data
Brief Title: Safety of Nintedanib in Real World in China
Status: Withdrawn | Type: Observational
Why Stopped: Company decision
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: China-Japan Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 1199-0412
Record Dates: First submitted 2022-12-22; First posted 2023-01-09 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis | interventions — nintedanib; pirfenidone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Nintedanib new users
  Interventions: Drug: nintedanib
- Pirfenidone new users
  Interventions: Drug: pirfenidone
- no drug-treated users: subjects who did not receive nintedanib, pirfenidone

INTERVENTIONS:
Drug: nintedanib — nintedanib
  Groups: Nintedanib new users
Drug: pirfenidone — pirfenidone
  Groups: Pirfenidone new users

SUMMARY:
The main objective of this study is to evaluate the incidence rates of adverse drug reactions (ADRs) and fatal adverse events (AEs) among idiopathic pulmonary fibrosis (IPF) patients in China who initiate nintedanib during the study period.

ELIGIBILITY:
Inclusion Criteria:

* Patients who initiate nintedanib during the study period
* Patients who initiate pirfenidone during the study period
* Patients who use neither nintedanib nor pirfenidone
* Patients who were diagnosed with IPF according to the 2011 American Thoracic Society (ATS)/European Respiratory Society (ERS)/Japanese Respiratory Society (JRS)/Latin American Thoracic Society (ALAT) guidelines in the past 3 months before recruitment
* Patients who are 40 years old and above when enrolled
* Patients who are willing to participate in the study and sign the informed consent form

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Idiopathic pulmonary fibrosis (IPF) patients in China:
  Patients who initiate nintedanib during the study (group 1). The index date for this group of patients is defined as the day when a patient initiates nintedanib; Patients who initiate pirfenidone during the study (group 2). The index date for this group of patients is defined as the day when a patient initiates pirfenidone; Patients who receive neither nintedanib nor pirfenidone (group 3). To define the index date for this group of patients, we will first calculate the average number of days between the first diagnosis of IPF and the day when nintedanib is initiated in group 1 patients (Xn). The index date for group 3 patients is defined as Xn days after the first diagnosis of IPF of a patient.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-12-29 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of adverse drug reactions (ADRs) during entire follow-up period | During entire follow-up period, up to 1 year
Incidence rate of adverse drug reactions (ADRs) during the 1-year follow-up period after the index date | During follow-up period after index date, up to 1 year
Incidence rate of fatal adverse events (AEs) during entire follow-up period | During entire follow-up period, up to 1 year
Incidence rate of fatal adverse events (AEs) during the 1-year follow-up period after the index date | During follow-up period after index date, up to 1 year

SECONDARY OUTCOMES:
Mean age at baseline of idiopathic pulmonary disease (IPF) patients in China who are new users of nintedanib, new users of pirfenidone, and those who receive neither of the two antifibrotic drug | At baseline
Percentage of each gender of idiopathic pulmonary disease (IPF) patients in China who are new users of nintedanib, new users of pirfenidone, and those who receive neither of the two antifibrotic drug | At baseline

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Link to PORTRAY study on clinicaltrials.gov — https://clinicaltrials.gov/ct2/show/NCT03666234?term=NCT03666234&draw=2&rank=1